CLINICAL TRIAL: NCT00934817
Title: An Open, Randomized, Two-Treatment, Crossover Study to Assess the Dose Proportionality of Glimepiride Between Amaryl M 1mg/500mg and 2mg/500mg (Glimepiride-Metformin Fixed Dose Combination Tablet) in Healthy Subjects
Brief Title: Dose Proportionality Study Comparing Amaryl-M 1/500 mg and Amaryl-M 2/500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Hye Jin Cheong / Head of Clinical Research Operation, Handok Pharmaceuticals, Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLIME_L_02279
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Volunteer
MeSH Terms: interventions — glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR sequential group (Experimental): Amaryl-M 1/500 mg in period 1, Amaryl-M 2/500 mg in period 2
  Interventions: Drug: Amaryl-M 2/500 mg; Drug: Amaryl-M 1/500 mg
- RT sequential group (Active Comparator): Amaryl-M 2/500 mg in period 1, Amaryl-M 1/500 mg in period 2
  Interventions: Drug: Amaryl-M 2/500 mg; Drug: Amaryl-M 1/500 mg

INTERVENTIONS:
Drug: Amaryl-M 2/500 mg — single oral administration in period 2 for TR sequential group, and in period 1 for RT sequential group, respectively
  Other Names: glimepiride 2 mg & metformin HCl 500 mg
Drug: Amaryl-M 1/500 mg — single oral administration in period 1 for TR sequential group, and in period 2 for RT sequential group, respectively
  Other Names: glimepiride 1 mg & metformin HCl 500 mg

SUMMARY:
The pharmacokinetics of glimepiride and metformin HCl will be compared after single dose intake of both combinations in order to answer the following questions:

* Is Amaryl-M 1/500 mg (Test tablet) proportional to Amaryl-M 2/500 mg tablet with regard to the glimepiride component?
* Is Amaryl-M 1/500 mg (Test tablet) tolerable comparing with Amaryl-M 2/500 mg?

DETAILED DESCRIPTION:
16 subjects were randomized to each of 2 sequence groups which have different treatment order of the study drug in each period.

Only healthy volunteers had screening tests such as medical inquiry, physical examination, clinical laboratory test, etc. within 4 weeks (-28d ~ -1d) prior to drug administration (1d) and those determined eligible for this study were selected and randomized between screening and 1 day prior to the first administration of study medication (-1d). Then, the subjects were admitted to the clinical research center of Seoul National University Hospital by 9 p.m. of -1d and then, they were not allowed to take anything except water.

After one week of washout period, subjects went on to the second phase of treatment period and were administered according to the treatment order in a crossover way. For the subjects who completed the study, post-study visit tests were performed after a designated time had passed.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 19 to 45 years of age, inclusive (age based on the date to give the informed consent)
* Ideal body weight (Broca index): between 50 to 90 kg, inclusive, and within ±20 % of Ideal Body Weight, [(Height in cm-100)×0.9]
* Subjects who are appropriate to participate in this study judged from clinical laboratory and physical examinations taken within 4weeks prior to the start of study
* Subjects who are able to abstain from caffeine or caffeine-containing products (e.g., coffee, cola, tea, chocolate), grapefruit and grapefruit containing products, alcohol and smoking within 7 days before dosing and during the hospitalization
* Subjects who give their informed consent voluntarily to participate in the study

Exclusion Criteria:

* History of allergies including drug allergy, except untreated, asymptomatic, seasonal allergies at the time of dosing
* Use any medication not considered acceptable by the clinical investigator during the last 10 days period before the start day of the study
* Use of any inducer or inhibitors of metabolizing enzymes during the last 28 days before the start day of the study.
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History of a significant surgical resection of gastrointestinal tract except appendectomy
* Abnormal clinical laboratory findings, especially for AST or ALT > 1.25 fold, total bilirubin > 1.5 fold of upper normal level
* Pregnant or lactating woman or woman of childbearing potential without medically acceptable birth control during the study
* Evidence of alcohol abuse (defined as regular alcohol intake that exceeds 24 oz [675 ml] of beer, 12 oz [340 ml] of wine or 160 ml of soju or 3 oz [85 ml] hard liquor per day [e.g., brandy, whiskey, gin]) or drug abuse
* Heavy smokers (> 10 cigarettes per day), or can't quit smoking during hospitalization
* Participation in clinical trials of any drug within 3 months prior to the start of study
* Donation of 200ml of whole blood within 4 weeks or 400ml within 12 weeks prior to the start of study
* Positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or HIV antibody
* Judged to be inappropriate for the study by the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentrations of glimepiride and metformin, PK parameters: AUCt, AUCinf, Cmax, Tmax, T1/2 | pre-dose (= 1d 0h), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 30 hrs after drug administration

SECONDARY OUTCOMES:
Physical examination, clinical laboratory tests | Screening, 2 day, 9 day, 13-15 day
Vital sign | screening, 1 day, 2 day, 8 day, 9 day, 13-15 day
Adverse event | 1 day, 2 day, 8 day, 9 day, 13-15 day

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Professor, Principal Investigator — Seoul National University Hospital